CLINICAL TRIAL: NCT05247034
Title: Evaluation of the Effect of Cocoa Supplementation on Biochemical and Clinical Profile and Sensory-motor Processing of Peripheral and Autonomic Diabetic Neuropathy: Randomized Clinical Trial
Brief Title: Effect of Cocoa Supplementation Peripheral and Autonomic Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Rebeca Kababie Ameo, Sponsor-Investigator, Anahuac University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202103; 202094 (Registry Identifier: Universidad Anáhuac México Norte)
Record Dates: First submitted 2022-01-05; First posted 2022-02-18 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Neuropathies
Keywords: Cocoa; Diabetic neuropathy; H-reflex; Cardiometabolic risk factor; Polyphenols; Antioxidants
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Diet for patients with diabetes + 4 capsules of cocoa powder, 500 mg each, daily for 12 weeks.
  Interventions: Dietary Supplement: Cocoa
- Control group (Placebo Comparator): Diet for patients with diabetes + 4 capsules of methylcellulose 500 mg each, daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cocoa — Each capsule of cocoa powder contains 12.5 mg of flavonoids, providing a total of 50 mg per day.
  Arms: Intervention group
Other: Placebo — Each capsule contains 500 mg of methylcellulose
  Arms: Control group

SUMMARY:
Type 2 diabetes mellitus is a high incidence disease in Mexico and is associated with the development of chronic degenerative complications such as diabetic neuropathy. The latter manifests itself as a set of disorders that occur as a consequence of a chronic hyperglycemic state that can induce oxidative stress and inflammation, resulting in damage to the autonomic and peripheral nervous system. In Mexico, it has been reported that this complication usually occurs between 29% and 90% of patients with diabetes.

Cocoa is a food with a high content of flavonoids, which are phenolic compounds with antioxidant and anti-inflammatory effects. Additionally, its consumption has been associated with a decrease in hyperglycemia and insulin resistance, improvement in mitochondrial function, and, based on the above, an effect on diabetic complications has been suggested; This has been demonstrated in in vivo and in vitro models, but not in the human population.

Once the symptoms of diabetic neuropathy have started, palliative treatments are prescribed, and to date there are no pharmacological compounds that have been shown to reverse the consequences of diabetic peripheral and autonomic neuropathy. Additionally, clinical trials of compounds with antioxidant properties have only performed subjective evaluations based on questionnaires on the perception of the improvement of diabetic neuropathy and some biochemical markers or nerve conduction tests, however, the results shown have not been conclusive.

This is why a double-blind, randomized controlled clinical trial is proposed, with the objective of evaluating the effect of cocoa supplementation in patients with type 2 diabetes mellitus and peripheral and autonomic diabetic neuropathy on a) the biochemical profile, which includes the evaluation of the glycemic and lipid profile, quantification of pro-inflammatory cytokines and oxidative stress markers; b) the clinical profile through the application of standardized questionnaires, anthropometric measurements and blood pressure, and c) somatosensory processing through the paired pulse H reflex test.

The hypothesis of this study is that cocoa supplementation will have a beneficial effect on the biochemical and clinical profile and somatosensory processing of peripheral and autonomic diabetic neuropathy.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a high incidence disease in Mexico and is associated with the development of chronic degenerative complications such as diabetic neuropathy. The latter manifests itself as a set of disorders that occur as a consequence of a chronic hyperglycemic state that can induce oxidative stress and inflammation, resulting in damage to the autonomic and peripheral nervous system. In Mexico, it has been reported that this complication usually occurs between 29% and 90% of patients with diabetes.

Cocoa is a food with a high content of flavonoids, which are phenolic compounds with antioxidant and anti-inflammatory effects. Additionally, its consumption has been associated with a decrease in hyperglycemia and insulin resistance, improvement in mitochondrial function, and, based on the above, an effect on diabetic complications has been suggested; This has been demonstrated in in vivo and in vitro models, but not in the human population.

Once the symptoms of diabetic neuropathy have started, palliative treatments are prescribed, and to date there are no pharmacological compounds that have been shown to reverse the consequences of diabetic peripheral and autonomic neuropathy. Additionally, clinical trials of compounds with antioxidant properties have only performed subjective evaluations based on questionnaires on the perception of the improvement of diabetic neuropathy and some biochemical markers or nerve conduction tests, however, the results shown have not been conclusive.

This is why a double-blind, randomized controlled clinical trial is proposed, with the objective of evaluating the effect of cocoa supplementation in patients with type 2 diabetes mellitus and peripheral and autonomic diabetic neuropathy on a) the biochemical profile, which includes the evaluation of the glycemic and lipid profile, quantification of pro-inflammatory cytokines and oxidative stress markers; b) the clinical profile through the application of standardized questionnaires, anthropometric measurements and blood pressure, and c) somatosensory processing through the paired pulse H reflex test. Hypothesis: The hypothesis of this study is that cocoa supplementation will have a beneficial effect on the biochemical and clinical profile and somatosensory processing of peripheral and autonomic diabetic neuropathy. Statistical analysis: For the evaluation of the intragroup variables, a statistical analysis will be carried out with ANOVA for repeated samples with Tukey's post hoc, or, where appropriate, Friedman with Dunn's post hoc, as well as Student's t for dependent groups, or in its case, with Wilcoxon. The intergroup comparison will be made with Student's T for independent samples, or if applicable, with Mann Whitney's U, considering p <0.05 as statistical significance and using the statistical software GraphPad Prism version 5.

The H reflex test will be performed by electrical stimulation through disposable surface electrodes connected to a constant current bipolar electrical stimulator (Digitimer DS8R). The recording of the electrophysiological signals will be carried out using surface electrodes connected to the signal acquisition and amplification system (LabChart and PowerLab 8/35, ADInstruments). The signals obtained will be sampled at 10 kilohertz (KHz) with a 0.5- 500 Hz band-pass filter. The signals will be stored in a computer for later analysis.

The placement of electrodes for stimulation will be carried out as follows: the active electrode (anode) at the level of the Achilles tendon, the positive electrode (cathode) above the inverted "v" between the calf muscles (gastrocnemius). Subsequently, the reference electrode will be placed at the level of the gastrocnemius heads. It will be stimulated behind the knee where the tibial nerve has its anatomical path.

The test will start with an intensity of 0 milliamp (mA) and then pulses will be given every 0.5 millivolts (mV) until the evoked potential (H reflex) is observed in a consistent and clearly identifiable way as a function of latency (35-45 ms). The electrical stimulus consists of the application of 1 square pulse (1 ms duration each pulse) every 10 seconds (10 pulses in total). The maximum intensity of the applied current will be according to the sensitivity and tolerance of the individual in both lower limbs during the tests on the sensory and motor nerves. The applied electrical pulse should not cause a painful sensation, but it can cause a tingling sensation. The test will be suspended if the individual reports pain or does not wish to continue with the research protocol. The "H" reflex test will be done in two parts. The first part of the protocol consists of determining the stimulus intensity vs. amplitude of motor responses from the appearance of the "M" wave and the "H" wave, for which the electric current will be increased in steps of 0.5 µA until the appearance of the waves. For this part, only one electrical pulse (1 ms duration) will be given every 10 seconds. The intensity of electrical current that will be used for the second part of the protocol will be that whose value in the amplitude curve of the H wave-electrical current intensity reaches 60% of the maximum amplitude. This stimulation value guarantees the reproducibility and minimum variability of this wave, which also prevents muscle contraction that contaminates the electrical register. The second part constitutes the paired electrical stimulation test in which two electrical pulses (1 ms in duration) will be produced at different frequencies between the pulses: 0.1, 1, 5 and 10 Hz. The interval between the paired pulses will be 10 s, until completing 10 series.

The electrophysiological recordings will be analyzed with the Clampfit 10.0 software. The latency and amplitude of the evoked potentials H1 and H2 will be determined for each electrical pulse and at all stimulation frequencies, taking the stimulus artifact as a reference. Subsequently, the ratio of the amplitude of the paired H2/H1 pulses will be determined to establish the modulation of spinal excitability. A ratio ≥0.6 for any stimulation frequency will be considered as an indicator of dysfunction in somatosensory processing according to Marshall et al.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-60 years with a diagnosis of type 2 diabetes mellitus and diabetic neuropathy
* Minimum time of diagnosis of T2DM of 5 years
* Who have a Michigan Neuropathy Screening Instrument (MNSI) score ≥2
* Male and Female
* Have them sign the informed consent letter

Exclusion Criteria:

* Subjects who modify their pharmacological treatment during the study
* Subjects who do not attend one of the intermediate consultations

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Cuéllar-Ramos, PhD, Study Director — Anahuac University; Gabriela Gutiérrez-Salmeán, PhD, Study Director — Anahuac University
Locations (3):
- Mexico (3):
  - Universidad Anáhuac México Norte, Huixquilucan, State of Mexico
  - Centro de Especialidades del Riñón, Naucalpan, State of Mexico
  - Clínica de Medicina Familiar "Nueva Oxtotitlán" ISSSTE, Toluca, State of Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 20 | 19
Completed | 16 | 17
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Organizational problems when attending appointments | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (8.67) | 53.7 (6.34) | 53.7 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 10 | 7 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 20 | 19 | 39
Toronto Clinical Scoring System [Mean (Standard Deviation); unit: units on a scale] — Toronto Clinical Study System is a quantitative scoring system for evaluating the severity of peripheral diabetic neuropathy that evaluates symptoms, reflexes and sensitivity. The minimum score is 0 points and the maximum is 19. It is classified as follows: 0-5 points, no neuropathy; 6-8 points, mild; 9-11 points, moderate; and 12-19 points, severe. For the purposes of this study, the total score, that is, the sum of all units on the scale, is reported. This is that, the higher the score (19 points), greater the severity (no grades were established according to the severity of the neuropathy).
  units on a scale | 9.31 (3.98) | 6.89 (3.47) | 8.10 (3.88)

OUTCOME MEASURES:

1. Primary Outcome: Toronto Clinical Scoring System (TCSS)
Description: It is a system of clinical evaluations carried out by the researcher to identify peripheral neuropathy, assigning a score to symptomatology, reflexes and sensory tests.
  For the purposes of this study, the total score, i.e., the sum of all units on the scale, is reported. The minimum score that can be obtained is 0 points, while the maximum is 19 points. This means that the higher the score, the greater the severity (no grades were established based on the severity of the neuropathy).
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: We could not obtain the Toronto Clinical Scoring System from one subject in the intervention group.
  Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
Score on a scale
  Change from baseline at Week 12 | -2.63 (2.24) | -1.84 (2.77)
  Baseline total score | 9.31 (3.98) | 6.89 (3.47)
  Final total score | 6.68 (4.41) | 5.05 (2.91)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p = 0.0125, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Rate-dependent Depression of the H-reflex
Description: Rate-dependent depression (RDD) is a measure of change in amplitude of the Hoffman (H) reflex over consecutive stimulations. Rate-dependent depression is impaired after disinhibition of spinal sensory processing caused by spinal cord injury.
  For the purposes of this study, the ratio of the amplitude of the pulses Hn/H1 ≥ 0.5 for stimulation frequencies 1, 5 and 10 Hz, was considered as an indicator of dysfunction in somatosensory processing. In healthy subjects, the ratio of the amplitude of the pulses Hn/H1 is expected to be <0.5.
  Each subject received 5 pulses for each stimulation frequency, and the average for each subject was determined. The group average was then obtained for each stimulation frequency (1, 5, and 10 Hz).
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: H reflex was found only in 8 subjects of the intervention group and in 10 subjects of the control group.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8 | 10
Ratio
  Change from baseline at Week 12 for 1 Hz | 0.13 (0.36) | 0.01 (0.28)
  Baseline 1 Hz mean: number analyzed (Participants) | 7 | 8
  Baseline 1 Hz mean | 0.87 (0.35) | 0.88 (0.33)
  Final 1 Hz mean | 0.99 (0.28) | 0.89 (0.16)
  Change from baseline at Week 12 for 5 Hz | -0.02 (0.51) | -0.03 (0.30)
  Baseline 5 Hz mean: number analyzed (Participants) | 8 | 8
  Baseline 5 Hz mean | 0.91 (0.67) | 0.71 (0.38)
  Final 5 Hz mean | 0.89 (0.21) | 0.65 (0.27)
  Change from baseline at Week 12 for 10 Hz | 0.13 (0.28) | -0.06 (0.20)
  Baseline 10 Hz mean: number analyzed (Participants) | 7 | 8
  Baseline 10 Hz mean | 0.56 (0.47) | 0.71 (0.42)
  Final 10 Hz mean | 0.72 (0.25) | 0.62 (0.30)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; For 1 Hz; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; 5 and 10 Hz; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Intervention Group; For 1, 5 and 10 Hz; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; For 1, 5 and 10 Hz; Test type: Other; p > 0.05, t-test, 2 sided

3. Secondary Outcome: BEST Questionnaire
Description: The questionnaire includes 4 questions that refer to gastrointestinal symptoms. This questions are measured in a scale from 1 (better health status) to 5 (worse health status) and it is related to gastrointestinal autonomic diabetic neuropathy.
  Final score: Minimum is 4 points (better health status) and maximum is 19 points (worse health status).
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale
  Change from baseline at Week 12 | -1.45 (2.62) | -2.21 (2.59)
  Baseline total score | 9.35 (2.75) | 9.05 (2.77)
  Final total score | 7.9 (2.67) | 6.84 (2.6)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p = 0.042, Friedman
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p = 0.015, Friedman

4. Secondary Outcome: Bristol Stool Form Scale
Description: It is composed of categories that include an image and an explanation, ranging from 1 to 7, being 1 separate hard pieces, which pass with difficulty and 7 watery stools. It is related to gastrointestinal autonomic diabetic neuropathy.
  The reported outcomes are the percentage of participants who had altered bristol stool form scale, that is, participants who were in categories 1, 2, 5, 6 and 7.
Time Frame: At baseline and 12 weeks
Population: Results presented are represented as percentage of subjects who had alteration in their bristol scale
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
percentage of participants
  Baseline altered bristol stool scale form | 40 | 57.8
  Final altered bristol stool scale form | 30 | 52.6
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p > 0.05, Z Test
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Z Test
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, Z Test

5. Secondary Outcome: Weight
Description: Weight of an individual in kg determined by the scale. The measurement is done without shoes and with as little clothing as possible. The subject must be placed in the center and remain still during the measurement.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: We could not obtain the weight measure from one participant of the intervention group.
  Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
kg
  Change from baseline at Week 12 | 0.38 (2.72) | -0.42 (2.18)
  Baseline | 73.5 (14.1) | 82.8 (13.8)
  Week 4 | 74.4 (14.8) | 82.5 (13.9)
  Week 8 | 74.1 (14.7) | 83 (13.7)
  Final | 73.8 (14.6) | 82.4 (13.9)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, ANOVA

6. Secondary Outcome: Waist Circumference
Description: Waist circumference in cm: The measuring tape is placed in a horizontal plane around the waist, taking the midaxillary line as a reference, locating the midpoint between the lower costal margin and the highest lateral border of the iliac crest.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
cm
  Change from baseline at Week 12 | -0.8 (2.19) | -1.38 (4.11)
  Baseline | 96.7 (7.49) | 103 (13.1)
  Week 4 | 96.5 (7.08) | 103 (11.7)
  Week 8 | 96 (7.33) | 103 (12)
  Final | 95.9 (7.28) | 102 (12)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, ANOVA

7. Secondary Outcome: Waist-to-Height Ratio
Description: It is obtained by dividing the waist circumference in cm by the height in cm, with a result of ≥ 0.5 indicating an increased risk for cardiometabolic disease.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: We could not obtain the height from 1 subject from the cocoa group. Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 19
Ratio
  Change from baseline at Week 12 | -0.00 (0.01) | -0.00 (0.02)
  Baseline | 0.6 (0.04) | 0.64 (0.09)
  Week 4 | 0.6 (0.04) | 0.64 (0.08)
  Week 8 | 0.6 (0.04) | 0.64 (0.09)
  Final | 0.6 (0.04) | 0.63 (0.09)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, ANOVA

8. Secondary Outcome: Abdominal Circumference
Description: Abdominal circumference in cm: The top of the hip bone and the top of the right iliac crest are located and the measuring tape is placed horizontally around the abdomen, at the level of the iliac crest, at the end of a normal expiration.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: Abdominal circumference couldn't be obtained from 2 subjects (1 from cocoa group and 1 from control group) Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 19 | 18
cm
  Change from baseline at Week 12 | -0.75 (2.45) | -1.02 (3.07)
  Baseline | 100 (9.31) | 106 (11.4)
  Week 4 | 100 (9.26) | 105 (11.7)
  Week 8 | 99.9 (9.27) | 105 (12)
  Final | 99.4 (9.01) | 104 (12.1)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, ANOVA

9. Secondary Outcome: Systolic Blood Pressure
Description: A sphygmomanometer is used to obtain blood pressure with the technique specified in the Clinical Practice Guidelines for the diagnosis and treatment of arterial hypertension at the first level of care, it is measured in mmHg.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
mmHg
  Change from baseline at Week 12 | -3.7 (11) | -3.78 (14.8)
  Baseline | 126 (14.6) | 127 (15.5)
  Week 4 | 125 (13.5) | 130 (17.2)
  Week 8 | 122 (12.2) | 125 (9.7)
  Final | 122 (14.2) | 124 (11.7)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, Friedman

10. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 9
Time Frame: At baseline, after 4, 8 and 12 weeks
Population: Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
mmHg
  Change from baseline at Week 12 | -2.32 (7.57) | -2.36 (10.1)
  Baseline | 79.9 (8.23) | 78.1 (7.98)
  Week 4 | 78.7 (8.78) | 79 (7.77)
  Week 8 | 79.8 (9.1) | 76.6 (7.13)
  Final | 77.6 (9.96) | 75.7 (7.97)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, Friedman

11. Secondary Outcome: Glucose
Description: Blood glucose concentration and is measured as mg/dL. For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
mg/dL
  Change from baseline at Week 12 | -17 (42.8) | -38.1 (55.9)
  Baseline mg/dL | 169 (62.6) | 195 (85.7)
  Final mg/dL | 152 (58.4) | 157 (63.6)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p = 0.0027, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Glycated Hemoglobin A1c
Description: Value of the fraction of hemoglobin that has glucose attached and is reported in percentage (%).
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
percentage of glycated hemoglobin
  Change from baseline at Week 12 | -0.17 (1.09) | -0.27 (0.60)
  Baseline % of glycated hemoglobin | 7.82 (1.9) | 8.28 (2.02)
  Final % of glycated hemoglobin | 7.72 (1.5) | 8 (2.04)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p = 0.0430, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Triglycerides
Description: Blood triglycerides concentration and is measured as mg/dL. For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
mg/dL
  Change from baseline at Week 12 | -4.96 (60.2) | -13.9 (44.6)
  Baseline mg/dL | 182 (81.4) | 179 (58.8)
  Final mg/dL | 177 (78.8) | 165 (52.1)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, t-test, 2 sided

14. Secondary Outcome: High-density Lipoprotein Cholesterol
Description: Blood high-density lipoprotein cholesterol concentration and is measured as mg/dL.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
mg/dL
  Change from baseline at Week 12 | -0.86 (3.71) | 2.18 (6.23)
  Baseline mg/dL | 37.8 (9.52) | 38.2 (9.12)
  Final mg/dL | 36.9 (7.5) | 40.4 (6.26)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Triglycerides/HDL Ratio
Description: It is obtained after dividing the serum concentration of triglycerides in mg/dL by the serum concentration of HDL in mg/dL. It does not have units.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
Ratio
  Change from baseline at Week 12 | -0.02 (1.98) | -0.74 (2.13)
  Baseline | 5.12 (2.84) | 4.99 (2.13)
  Final | 5.1 (2.9) | 4.25 (1.31)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, t-test, 2 sided

16. Secondary Outcome: Low-density Lipoprotein Cholesterol
Description: Blood low-density lipoprotein cholesterol concentration and is measured as mg/dL.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
mg/dL
  Change from baseline at Week 12 | 8.88 (22.1) | 4.15 (18.1)
  Baseline mg/dL | 112 (31.8) | 108 (31.3)
  Final mg/dL | 121 (35.2) | 112 (34.7)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, t-test, 2 sided

17. Secondary Outcome: Neutrophil/Lymphocyte Ratio
Description: It is obtained by dividing the serum concentration of the absolute number of neutrophils by the serum concentration of the absolute number of lymphocytes. Without unit.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
Ratio
  Change from baseline at Week 12 | -0.09 (0.77) | 0.15 (0.45)
  Baseline | 1.96 (0.86) | 1.76 (0.55)
  Final | 1.87 (1.07) | 1.92 (0.61)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, t-test, 2 sided

18. Secondary Outcome: Diabetes 39 Instrument
Description: It is a self-administered instrument that allows patients to describe how their QOL was affected during the previous month in five domains: energy and mobility (15 questions), diabetes control (12 questions), anxiety and worry (4 questions), social impact (5 questions), and sexual behavior (3 questions). Responses are scored on a seven-point scale that ranged from "not affected at all" (score = 1) to "extremely affected" (score = 7). All responses are summed and it is applied a linear transformation to a 0-100 scale. Lower scores indicated a better QOL.
  For the data represented in the row "Change from baseline at Week 12", it is the delta of the final measurement vs. the initial measurement, that is, the final measurement minus the baseline measurement.
Time Frame: At baseline and after 12 weeks
Population: Intention-to-treat analysis was performed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 19
score on a scale
  Change from baseline at Week 12 | -9.19 (11.6) | -5.26 (19)
  Baseline total score | 43.4 (26.8) | 35.6 (22.6)
  Final total score | 34.2 (25.8) | 30.4 (24.5)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Comparing row "Change from baseline at Week 12"; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Intervention Group; Test type: Other; p = 0.0007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control Group; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
Evaluation of inflammation and oxidative stress parameters was proposed, however, given the cost involved, neutrophil/lymphocyte ratio was used as a marker of inflammation, but oxidative stress was not measured.

It was necessary to include different centers for recruiting potential candidates.

The follow-up period was established based on human resources and the budget; however, it can be considered a short time to identify significant differences in outcomes such as RDD of the H-reflex.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT05247034/Prot_SAP_ICF_000.pdf